CLINICAL TRIAL: NCT00532558
Title: A Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of Lapaquistat Acetate 50 mg vs Placebo in Subjects With Hypercholesterolemia, With an Optional Open-Label Extension
Brief Title: Efficacy of Lapaquistat Acetate on Blood Cholesterol Levels in Treating Subjects With Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Overall profile of the compound does not offer significant clinical advantage to patients over currently available lipid lowering agents
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-475_306; U1111-1122-8417 (Registry Identifier: WHO)
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate 50 mg QD (Experimental)
  Interventions: Drug: Lapaquistat acetate
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lapaquistat acetate — Lapaquistat acetate 50 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 50 mg QD
Drug: Placebo — Lapaquistat acetate placebo-matching tablets, orally, once daily for up to 12 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of the study is to determine the reduction of LDL-cholesterol level after treatment with 50 mg per day of lapaquistat acetate once daily (QD).

DETAILED DESCRIPTION:
This study is being conducted to determine the potential of lapaquistat acetate 50 mg per day to lower LDL-C levels compared with placebo. This study is also being conducted to further evaluate the safety and tolerability of lapaquistat acetate 50 mg over a period of 12 weeks. An optional, 48-week, open-label extension will follow the 12 week, double-blind treatment period to evaluate the long-term safety and tolerability of lapaquistat acetate 50 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception from screening throughout the duration of the study and for 30 days following the last dose.
* Prior to Randomization, the participant has a mean low density lipoprotein cholesterol level greater than or equal to 130 mg/dL and less than or equal to 190 mg/dL for 2 consecutive samples.
* Prior to Randomization, the subject has mean triglyceride level greater than or equal to 400 mg/dL for 2 consecutive samples.
* Is willing and able to comply with the recommended, standardized diet.

Exclusion Criteria:

* Has an nine aminotransferase or aspartate aminotransferase level greater than 1.5 times the upper limit of normal, identified during screening.
* Has a serum creatinine greater than 133 mmol/L, identified during screening.
* Has a creatine kinase greater than 3 times the upper limit of normal, identified during screening.
* Has active liver disease or jaundice.
* Has taken any fibrates within 42 days of Visit 1 or any lipid-lowering therapy for at least 30 days prior to Screening.
* Has a previous history of cancer that has been in remission for less than 5 years prior to the first dose of study medication.
* Has an endocrine disorder, such as Cushing's syndrome, hyperthyroidism, or inappropriately treated hypothyroidism affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, unstable angina, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdominal aortic aneurysm, coronary angioplasty, coronary or peripheral arterial surgery, or multiple risk factors that confer a 10-year risk for cardiovascular heart disease greater than 20% based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen or hepatitis C virus antibody test, as determined by medical history.
* Has a positive human immunodeficiency virus status or is taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Has received any investigational medication 30 days prior to screening, (for drugs with a long half-life, within a period of less than 5 times the drug's half-life) or is participating in an investigational study.
* Has received lapaquistat acetate in a previous clinical study or as a therapeutic agent.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the specialized diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension
* Has had inflammatory bowel disease or any other malabsorption syndrome, or has had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of high alcohol intake within the previous 2 years.
* Has type 1 or 2 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in fasting plasma Low Density Lipoprotein cholesterol | Week 12 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Total Cholesterol | Week 12 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in apolipoprotein A1 Timeframe: Week 12 or Final Visit | Week 12 or Final Visit
Change from Baseline in apolipoprotein B | Week 12 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 12 or Final Visit
Change from Baseline in Triglycerides | Week 12 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (60):
- Estonia (2):
  - Tallinn
  - Tartu
- Hungary (6):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Érd
  - Pécs
  - Szekszárd
- Israel (8):
  - Beersheba
  - Hadera
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Safed
  - Tel Aviv
- Latvia (3):
  - Daugavpils
  - Kuldīga
  - Riga
- Netherlands (8):
  - Amsterdam
  - Breda
  - GA Nijmegen
  - Groningen
  - Hoorn
  - Rotterdam
  - Utrecht
  - Zoetermeer
- Norway (5):
  - Ålesund
  - Elverum
  - Hamar
  - Kongsberg
  - Oslo
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Saratov
  - Tyumen
  - Volgograd
- Slovakia (6):
  - Bratislava
  - Dolný Kubín
  - Košice
  - Nitra
  - Nové Mesto nad Váhom
  - Trebišov
- Spain (5):
  - Córdoba
  - Madrid
  - Pontevedra
  - REUS (Tarragona)
  - Valencia
- Ukraine (6):
  - Dnipro
  - Kharkiv
  - Kiev
  - Kyiv
  - Lutsk
  - Lviv
- United Kingdom (6):
  - Belfast
  - Bolton
  - Glasgow, Scotland
  - Oldham
  - Paignton, Devon
  - Sheffield